CLINICAL TRIAL: NCT00926016
Title: Assessment of the Efficacy of Pioglitazone on Viral Kinetics, Cytokines, and Innate Immunity in a Group of Insulin Resistant, Treatment Naïve, Chronic Hepatitis C, Genotype 1 Patients
Brief Title: Pioglitazone on Viral Kinetics, Cytokines and Innate Immunity in Insulin Resistant CHC GT 1 Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Collaborators: The Geneva Foundation (Other)
Responsible Party: Principal Investigator, Stephen A Harrison, Principal Investigator, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: C.2006.152
Record Dates: First submitted 2009-06-22; First posted 2009-06-23 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Chronic Hepatitis C
Keywords: Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pioglitazone (Active Comparator): Treatment with pioglitazone 45 mg a day for 3 months
  Interventions: Drug: Pioglitazone (Actos)
- No intervention (No Intervention): Monitoring period without pioglitazone for 3 months

INTERVENTIONS:
Drug: Pioglitazone (Actos) — pioglitazone 45 mg a day
  Arms: pioglitazone

SUMMARY:
The purpose of this study is to determine if rosiglitazone, a medicine used to treat diabetes, improves response to anti-viral treatment.

DETAILED DESCRIPTION:
The aim of the study will be to determine if an insulin sensitizing thiazolidinedione (TZD) improves (1) baseline viremia, (2) enhances viral kinetics, (3) improves cytokine profiles and (4) up regulates innate cellular immunity (presumably adaptive immunity is up regulated as well) as measured by the bioactivity of the collected biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* HCV-Ab or HCV-RNA by PCR Positive for at least six months (to rule out acute seroconversion)
* Serum positive for HCV-RNA by PCR assay
* Must have insulin resistance, defined as a QUICKI score < 0.35. QUICKI
* Liver biopsy consistent with CHC within 24 months prior to enrollment
* Compensated liver disease with the following minimum hematological, biochemical, and serologic criteria at the Screening Visit (WNL = within normal limits):

  * Hemoglobin values of >12 gm/dL for females and >13 gm/dL for males.
  * WBC >3,000/ mm3
  * Neutrophil count > 1,500/mm3
  * Platelets >65,000/ mm3
  * Direct bilirubin, within 20% of ULN
  * Indirect bilirubin, within normal limits (WNL)
  * Albumin >3gm/dL
  * Serum creatinine < 20% above the ULN
  * TSH WNL
  * Alpha fetoprotein value < 100 ng/mL

Exclusion Criteria:

* Prior interferon based therapy
* Use of insulin
* Fasting glucose levels > 200 mg/dl
* Women who are pregnant or breast-feeding
* No other thiazolidinedione after liver biopsy and/or during the entire study (
* Hepatitis C of non-genotype 1
* Suspected hypersensitivity to pioglitazone
* Any cause for liver disease other than chronic hepatitis C, insulin resistance, or NAFLD, including but not limited to:

  * Hemochromatosis
  * Alpha-1 antitrypsin deficiency
  * Co-infection with HBV
  * Wilson's disease
  * Autoimmune hepatitis
  * Significant alcohol use
  * Drug-related liver disease
* Any condition that would prevent the subject from having a liver biopsy.
* Hemoglobinopathies that could potentially compromise patient safety
* Evidence of advanced liver disease such as history or presence of ascites, bleeding varices, spontaneous encephalopathy.
* Participants with organ transplants other than cornea and hair transplant.
* Any known preexisting medical condition that could interfere with the subject's participation in and completion of the protocol such as:

  * Preexisting psychiatric condition, especially severe depression, or a history of severe psychiatric disorder, such as major psychoses, suicidal ideation and/or suicidal attempt are excluded
  * Substance abuse, such as alcohol, IV drugs and inhaled drugs
  * Alcohol consumption is to be strongly discouraged
  * Seizure disorders not controlled with medication
  * Significant cardiovascular dysfunction within the past 12 months
  * Chronic pulmonary disease with documented pulmonary hypertension
  * Immunologically mediated disease [e.g., inflammatory bowel disease (Crohn's disease, ulcerative colitis)], rheumatoid arthritis, idiopathic thrombocytopenia purpura, systemic lupus erythematosis, autoimmune hemolytic anemia, scleroderma, severe psoriasis, clinical cryoglobulinemia with vasculitis
* Any medical condition requiring, or likely to require, chronic systemic administration of steroids during the course of the study
* Evidence of an active or suspected cancer or a history of malignancy where the risk of reoccurrence is ≥ 20% within two years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-06; Primary Completion 2010-03 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Improvement in baseline viremia and viral kinetics, and/or pro-inflammatory cytokines decrease, and/or markers of innate immunity are upregulated to position a more favorable response to current CHC therapy. | 104 days

CONTACTS AND LOCATIONS:
Overall Officials: Stephen A Harrison, MD, Principal Investigator — Brooke Army Medical Center
Locations (1):
- Brooke Army Medical Center, San Antonio, Texas, United States